CLINICAL TRIAL: NCT02103114
Title: Double Blind Randomized Placebo-controlled Study in Children (<6mo) Comparing the Effects of Anti-thrombin III (ATIII) or Placebo on the Coagulation System in Infants With Known Low ATIII Levels Undergoing Open Congenital Cardiac Surgery
Brief Title: Anti-thrombin III (ATIII) vs Placebo in Children (<7mo) Undergoing Open Congenital Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00051186
Record Dates: First submitted 2014-04-01; First posted 2014-04-03 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: ATIII Deficiency
MeSH Terms: interventions — Antithrombin III

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anti-thrombin III (Experimental)
  Interventions: Drug: Anti-thrombin III
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Anti-thrombin III — Intraoperatively- (correcting to 100%) according to the following formula:
  Units required = ((100%- baseline ATIII level*%) X body weight)/1.4
  * expressed as a % normal level based on functional ATIII assay
  Other Names: Thrombate III
  Arms: Anti-thrombin III
Other: Placebo — Normal saline placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether the administration of ATIII during the intra-operative period results in improved anticoagulation for cardiopulmonary bypass (CPB) and an attenuation of the activation of the coagulation cascade, as represented by a decrease in fibrin degradation products. The investigators believe this benefit would extend into the post-operative period resulting in a decreased incidence of thrombosis generation, as represented by a decrease in fibrin degradation products in the ICU period.

DETAILED DESCRIPTION:
If Preoperative ATIII functional assay level is less than 70% patients would be enrolled and randomized to either Placebo (normal saline) or ATIII.

ELIGIBILITY:
Inclusion Criteria:

* All patients less than 7 months of age going for cardiac surgery that will require cardiopulmonary bypass (CPB) with a documented ATIII level below 70%

Exclusion Criteria:

* Less than 2.5kg
* Known or suspected hereditary ATIII deficiency (family history of venous thrombosis with decreased plasma levels of ATIII and no other potential causes of acquired decreased ATIII)
* On Ecmo (extracorporeal membrane oxygenation ) at time of surgery
* Known history of thrombosis
* Renal failure as described by the pediatric RIFLE criteria
* H/o intracranial hemorrhage
* Prematurity less than 37 weeks estimated gestational age
* Previously diagnosed pro-thrombotic or hemorrhagic disorder
* Prior ATIII supplementation
* Prior therapeutic anticoagulant use

Max Age: 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06-27 (Actual); Study Completion 2016-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Jooste, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five subjects enrolled but withdrew prior to randomization
Period: Overall Study
Arm/Group | Anti-thrombin III | Placebo
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-thrombin III | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: days] | 9.8 (19.7) | 17.2 (30.2) | 14.6 (26.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Mean and Standard Deviation (SD) of the Calibrated Automated Thrombography (CAT) Measurements of the Control and ATIII Groups at Time 5 (on Arrival in ICU)
Description: Evidence of decreased activation of the coagulation and fibrinolytic systems represented by a difference in the mean and Standard Deviation (SD) of the Calibrated Automated Thrombography (CAT) measurements of the control and ATIII groups at Time 5 (on arrival in ICU).
Time Frame: Time 5 (on arrival in ICU)
Population: The laboratory was unable to perform this blood assay due to technical issues and no results were generated.
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Difference in the Mean and SD of the Calibrated Automated Thrombography (CAT) Measurements of the Control and ATIII Groups at Times 5-Time 7 (ICU Arrival to Post Operative Day 4)
Description: Evidence of decreased activation of the coagulation and fibrinolytic systems represented by a difference in the mean and SD of the Calibrated Automated Thrombography (CAT) measurements of the control and ATIII groups at times 5-Time 7 (ICU arrival to Post Operative Day 4)
Time Frame: ICU arrival (Time 5) to Time 7 (Post-operative Day 4)
Population: The laboratory was unable to perform this blood assay due to technical difficulties and no results were generated.
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Difference in the Mean the ATIII (Functional Assay) of the Control and ATIII Groups at T1, T2, T3, T5, T6 and T7
Description: Evidence of decreased activation of the coagulation and fibrinolytic systems represented by a difference in the mean of the ATIII (functional assay) of the control and ATIII groups at T1, T2, T3, T5, T6 and T7 (Baseline, 30 min after study drug, 30 min on CPB, Arrival in ICU, POD 2, and POD 4). Data reported as % Functional Activity, which is calculated as the ability of Antithrombin (AT) to suppress FIIa or FXa in the presence of heparin compared to normograms, and expressed as a percentage.
Time Frame: T1, T2, T3, T5, T6 and T7
Measure: Mean (Standard Deviation); unit: % Functional Activity
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
% Functional Activity
  T1 (Baseline) | 54 (12) | 54 (13)
  T2 (30 minutes post study drug) | 99 (19) | 49 (16)
  T3 (30 minutes on CPB) | 83 (20) | 55 (27)
  T5 (Arrival in ICU) | 82 (18) | 63 (19)
  T6 (POD 2) | 58 (15) | 57 (14)
  T7 (POD 4) | 70.7 (20) | 66 (17)
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T1 (Baseline); p = 0.982, t-test, 2 sided
Statistical Analysis 2: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T2 (30 minutes after study drug); p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T3 (30 minutes on CPB); p = 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T5 (Arrival in ICU); p = 0.003, t-test, 2 sided
Statistical Analysis 5: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T6 (POD 2); p = 0.840, t-test, 2 sided
Statistical Analysis 6: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T7 (POD 4); p = 0.475, t-test, 2 sided

4. Secondary Outcome: Difference in the Median of the ATIII (Functional Assay) of the Control and ATIII Groups at T4
Description: Evidence of decreased activation of the coagulation and fibrinolytic systems represented by a difference in the median of the ATIII (functional assay) of the control and ATIII groups at T4 (just prior to coming off of CPB). Data reported as % Functional Activity, which is calculated as the ability of Antithrombin (AT) to suppress FIIa or FXa in the presence of heparin compared to normograms, and expressed as a percentage.
Time Frame: T4 (just prior to coming off of CPB)
Measure: Median (Inter-Quartile Range); unit: % Functional Activity
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
% Functional Activity | 78.0 [69.5 to 95.0] | 69.0 [35.0 to 89.0]
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T4 (just prior to coming off of CPB); p = 0.048, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Difference in the Median of the D Dimer of the Control and ATIII Groups at T1, T5, T6 and T7
Description: Evidence of decreased activation of the coagulation and fibrinolytic systems represented by a difference in the median of the D dimer of the control and ATIII groups at T1 (Baseline), T5 (Arrival in Intensive Care Unit), T6 (Post-Operative Day 2) and T7 (Post-Operative Day 4).
Time Frame: T1, T5, T6 and T7
Measure: Median (Inter-Quartile Range); unit: mcg/ml
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
mcg/ml
  T1 (Baseline) | 1.1 [0.7 to 1.5] | 0.9 [0.7 to 1.9]
  T5 (Arrival in ICU) | 0.6 [0.5 to 0.9] | 1.0 [0.6 to 1.5]
  T6 (POD 2) | 1.3 [0.9 to 2.0] | 1.7 [1.0 to 2.9]
  T7 (POD 4) | 3.2 [2.5 to 4.3] | 5.6 [4.3 to 8.4]
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T1 (Baseline); p = 0.855, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T5 (Arrival in ICU); p = 0.225, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T6 (POD 2); p = 0.313, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T7 (POD 4); p = 0.008, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Residual Heparin at the ICU Arrival Time Point Represented by a Decreased Anti Factor Xa Level.
Description: Evidence of a decreased amount of residual heparin at the Intensive Care Unit arrival time point (T5) represented by a decreased anti factor Xa level.
Time Frame: T5 (Intensive Care Unit Arrival)
Population: In both arms, heparin level was undetectable as Anti factor Xa level was less than or equal to 0.1 IU/ml in all subjects.
Measure: Mean (Standard Deviation); unit: International Units/milliter
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
International Units/milliter | 0.1 (0) | 0.1 (0)

7. Secondary Outcome: Evidence of Decreased Inflammation Represented by a Decrease in Inflammatory Markers in the ATIII Group
Description: Evidence of decreased inflammation represented by a decrease in inflammatory markers in the ATIII group.
Time Frame: Baseline (T1) to Post-Operative Day 4 (T7)
Population: Laboratory testing not performed.
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Total Dose of Heparin While on Cardiopulmonary Bypass
Description: Total dose of Heparin while on Cardiopulmonary Bypass
Time Frame: T1 (Baseline) to T5 (Arrival in ICU)
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
units | 3775 [3400.0 to 5700.0] | 5000 [4200.0 to 6300.0]
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T1 (Baseline) to T5 (Arrival in ICU); p = 0.056, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Protamine Dose Determined by Hemostasis Management System Machine (mg/kg)
Description: Protamine dose determined by Hemostasis Management system machine (mg/kg)
Time Frame: T1 (Baseline) to T5 (Arrival in ICU)
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
mg/kg | 9.8 [9.1 to 10.1] | 10.0 [6.5 to 10.7]
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — T1 (Baseline) to T5 (Arrival in ICU); p = 0.545, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Total Volume of Blood Products While on CPB
Description: Total volume of blood products exposed intraoperatively including the pump prime (ml/kg)
Time Frame: Baseline (intraoperatively) (Time 1) to before termination of bypass (Time 4)
Measure: Mean (Standard Deviation); unit: mls
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
mls
  Total Volume Red Blood Cells | 57 (103.9) | 101.5 (128.9)
  Total Volume Fresh Frozen Plasma | 68.5 (121.5) | 141.9 (133.6)
  Total volume ultrafiltration Platelet transfusion | 89.7 (44.2) | 72.6 (54)
  Total volume Cryoprecipitate transfusion | 35.4 (22.8) | 33.8 (32.5)

11. Secondary Outcome: Time From Protamine Administration to Skin Dressing
Description: Time from protamine administration to skin dressing
Time Frame: Baseline (intraoperatively) (Time 1) to before termination of bypass (Time 4)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
minutes | 107.0 [65.0 to 123.0] | 89.0 [60.0 to 155.0]
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — Baseline (intraoperatively) (Time 1) to before termination of bypass (Time 4); p = 0.757, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Total Volume of Fresh Frozen Plasma Given Prior to CPB
Description: Total volume of Fresh Frozen Plasma given prior to CPB, including the pump prime (ml/kg)
Time Frame: Baseline (intraoperatively) (Time 1) to before termination of bypass (Time 4)
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
ml/kg | 15 (67.1) | 5.8 (25.5)

13. Secondary Outcome: Incidence of Recombinant Factor 7a (VIIa) Use Intraoperatively
Description: Incidence of Recombinant Factor 7a (VIIa) Use Intraoperatively
Time Frame: Baseline (Intraoperatively)
Measure: Number; unit: count of participants
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
count of participants | 5 | 5

14. Secondary Outcome: Volume of Postoperative Blood Loss
Description: Volume of postoperative blood loss from 10min post protamine administration to 24 hour post protamine administration- (ml/kg)
Time Frame: From 10min post protamine administration to 24 hour post protamine administration
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
ml/kg
  24 hour postop Fresh Frozen Plasma exposures | 0.8 (3.4) | 2.8 (7.3)
  24 hour postop Platelet exposures | 0 (0) | 2.7 (5.6)
  24 hour postop Cryoprecipitate exposures | 0 (0) | 2.1 (5.4)
  24 hour postop Red Blood Cell exposures | 3.9 (7.3) | 10.1 (16.4)
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 0.2741, t-test, 2 sided; 24 hour postop Fresh Frozen Plasma exposures
Statistical Analysis 2: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 0.0351, t-test, 2 sided; 24 hour postop Platelet exposures
Statistical Analysis 3: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 0.073, t-test, 2 sided; 24 hour postop Cryoprecipitate exposures
Statistical Analysis 4: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 0.0196, t-test, 2 sided; 24 hour postop Red Blood Cell exposures

15. Secondary Outcome: Chest Tube Output (Protamine Time Plus 24 Hours) in Milliliters
Description: Chest Tube output (protamine time plus 24 hours) in milliliters
Time Frame: protamine time plus 24 hours
Measure: Median (Inter-Quartile Range); unit: milliters
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
milliters | 59.0 [46.5 to 83.5] | 113.0 [67.0 to 210.0]
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — protamine time plus 24 hours; p = 0.016, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Number of Total Blood Product Units Transfused by Type 24-hours Post-operatively by Group
Description: Number of packed Fresh frozen plasma units, Platelet Units, cryo-precipitate units, and Red Blood Cell units transfused 24 hours post-operatively for each group (not total units transfused for each subject)
Time Frame: 24 Hours Post-Operatively
Population: Unable to be calculated accurately as blood products given in CPB prime were only designated in Units administered and not mls (no record of how many mls present in each unit). Therefore unable to back calculate total mls given from start of surgery to 24 hours postop
Measure: Number; unit: Units
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
Units
  Fresh Frozen Plasma Units | 1 | 3
  Platelet Units | 0 | 4
  Cryo-Precipitate Units | 0 | 3
  Red Blood Cell Units | 5 | 9

17. Secondary Outcome: Number of Total Blood Product Units Transfused 24-hours Post-operatively by Group
Description: Number of total blood product units (including packed Fresh frozen plasma units, Platelet Units, cryo-precipitate units, and Red Blood Cell units) transfused 24 hours post-operatively for each group (not total units transfused for each subject)
Time Frame: 24 Hours Post-Operatively
Measure: Number; unit: Units
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
Units | 6 | 19
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Equivalence — 24 Hours Post-Operatively; p = 0.0004, Fisher Exact

18. Secondary Outcome: Total Dose of Recombinant Factor 7a (VIIa) Used Intraoperatively
Description: Total Dose of rescue recombinant factor 7a (VIIa) used intraoperatively
Time Frame: Intraoperatively
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
mcg | 56.1 (118.2) | 70.6 (174.1)
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 0.927, t-test, 2 sided

19. Secondary Outcome: Length of Post Operative Ventilation in Days
Description: Length of post operative ventilation in days
Time Frame: ICU arrival (Time 5) to Time 7 (Post-Operative Day 4)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
days | 3.9 (2) | 3.6 (1.3)
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 0.738, t-test, 2 sided

20. Secondary Outcome: Incidence of Extracorporeal Membrane Oxygenation (ECMO) Support Within 24 Hours Postoperatively
Description: Study the safety profile of dosing the ATIII by monitoring the incidence of extracorporeal membrane oxygenation (ECMO) support within 24 hours postoperatively.
Time Frame: Baseline (intraoperatively) (Time 1) to Time 7 (Post OP Day 4)
Measure: Number; unit: number
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
number | 0 | 2
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 0.231, Fisher Exact

21. Secondary Outcome: Incidence of Mediastinal Exploration Within 24 Hours Postoperatively
Description: Study the safety profile of dosing the ATIII by monitoring the incidence of mediastinal exploration within 24 hours postoperatively
Time Frame: Baseline (intraoperatively) (Time 1) to Time 7 (Post OP Day 4)
Measure: Number; unit: count of participants
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
count of participants | 2 | 3
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 0.661, Fisher Exact

22. Secondary Outcome: Incidence (Number) of Thrombotic Events Documented
Description: Study the safety profile of dosing the ATIII by monitoring the incidence (number) of thrombotic events documented.
Time Frame: Baseline (intraoperatively) (Time 1) to Time 7 (Post OP Day 4)
Measure: Number; unit: events
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
events | 0 | 0

23. Secondary Outcome: Incidence of New Onset Renal Failure, Defined by Stage 3 of the AKIN Criteria
Description: Study the safety profile of dosing the ATIII by monitoring the incidence of new onset renal failure, defined by stage 3 of the Acute Kidney Injury Network (AKIN) criteria.
  1. Serum creatinine increase ≥26.5 μmol/l (≥0.3 mg/dl) or increase to 1.5-2.0-fold from baseline, urine output <0.5 ml/kg/h for 6 hours
  2. Serum creatinine increase >2.0-3.0-fold from baseline, urine output <0.5 ml/kg/h for 12 hours
  3. Serum creatinine increase >3.0-fold from baseline or serum creatinine ≥354 μmol/l (≥4.0 mg/dl) with an acute increase of at least 44 μmol/l (0.5 mg/dl) or need for Renal replacement therapy (RRT), urine output <0.3 ml/kg/h for 24 h or anuria for 12 hours or need for RRT
Time Frame: Baseline (intraoperatively) (Time 1) to Time 7 (Post OP Day 4)
Measure: Number; unit: count of participants
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
count of participants | 1 | 1
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 1.0, Fisher Exact

24. Secondary Outcome: Incidence (Number) of Newly Diagnosed Intracranial Hemorrhage
Description: Study the safety profile of dosing the ATIII by monitoring the incidence (number) of newly diagnosed intracranial hemorrhage
Time Frame: Baseline (intraoperatively) (Time 1) to Time 7 (Post OP Day 4)
Measure: Number; unit: participants
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
participants | 1 | 3
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 0.342, Fisher Exact

25. Secondary Outcome: Length of Time to Delayed Sternal Closure Measured in Days
Description: Study the safety profile of dosing the ATIII by monitoring the length of time to delayed sternal closure measured in days
Time Frame: Baseline (intraoperatively) (Time 1) to Time 7 (Post OP Day 4)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Anti-thrombin III | Placebo
Number analyzed (Participants) | 20 | 19
days | 2.7 (2.1) | 2.7 (2.2)
Statistical Analysis 1: Comparison: Anti-thrombin III vs Placebo; Test type: Superiority or Other; p = 0.961, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline (intraoperatively) until post-operative day four.
Arm/Group | Anti-thrombin III | Placebo
Serious Adverse Events (participants affected / at risk) | 3/20 | 8/20
Other Adverse Events (participants affected / at risk) | 3/20 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-thrombin III (N=20) | Placebo (N=20)
Hypotension R/T chest fluid retention (not bleeding) (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Right-sided tonic clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension R/T bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Shock (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Right-sided subdural hematoma (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhage (Surgical and medical procedures) | 1 (1) | 1 (1)
Bradycardia (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Surgical and medical procedures) | 1 (1) | 0 (0)
ECMO (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intraop Bleeding (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-thrombin III (N=20) | Placebo (N=20)
Junctional ectopic tachycardia (Cardiac disorders) | 1 | 0
Junctional rhythm tachycardia (Cardiac disorders) | 0 | 1
Hematochezia (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Low Hematocrit (Blood and lymphatic system disorders) | 1 | 0
Desaturation (Blood and lymphatic system disorders) | 0 | 1
Intermittent PVCs R/T Low K, Low Mg (Blood and lymphatic system disorders) | 0 | 1
SVTs (Cardiac disorders) | 0 | 1
Echogenic focus in occipital parietal region (Nervous system disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Hemoparitoneum (Blood and lymphatic system disorders) | 0 | 1
Posterior subdural hematoma (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Right Lung Collapse (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes